CLINICAL TRIAL: NCT01717339
Title: Sleep Apnea and Vascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Virend Somers, PI, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 12-006285
Record Dates: First submitted 2012-10-25; First posted 2012-10-30 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: OSA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal Subjects (Other): Non-OSA (Obstructive sleep apnea) patients
  Interventions: Other: Sleep Study
- OSA subjects (Other): (Obstructive sleep apnea) OSA subjects
  Interventions: Other: Sleep Study

INTERVENTIONS:
Other: Sleep Study

SUMMARY:
Obstructive sleep apnea (OSA) is associated with endothelial dysfunction and the development of cardiovascular disease. It is unclear how OSA results in endothelial dysfunction, but given the association between OSA and obesity, adipose-derived hormones (adipokines) are likely to be involved. Leptin, an adipokine upregulated in patients with OSA, has been shown to be associated with deleterious effects on vascular function resulting in impaired endothelial function. This proposal is directed at investigating the molecular mechanisms of endothelial dysfunction in OSA patients. We hypothesize that endothelial dysfunction associated with OSA is a result of molecular alterations within endothelial cells. As a part of these studies we will look at NO signaling pathways in adipose tissue and microvessels from normal and OSA subjects.

ELIGIBILITY:
Inclusion Criteria:

* Non OSA, and newly diagnosed OSA subjects, naïve to CPAP treatment, aged 18-65 years, with BMI less than or equal to 55 kg/m2, who are free of all chronic diseases including diabetes, and cardiovascular diseases, will be recruited for our study. Subjects with dyslipidemia and hypertension will be allowed to participate in the study. Subjects taking anti-depressents, and anithypertensives will be allowed to participate in the study. Also, subjects taking beta blockers and beta agonists will be allowed to participate in the study.

If a subject is on aspirin or any other anti-inflammatory medication but free of known vascular disease and depending on the indication, the study doctor may ask the subject to suspend aspirin or anti-inflammatory therapy for 7 days prior to participation in the study. In the event that the subjects does not stop the aspirin or other anti-inflammatory medication, they will not be able to participate in the study because of the risk of bleeding during the fat biopsy.

Exclusion Criteria:

* Body weight >450 pounds (204.5kg)
* Pregnancy.
* Anemic (hemoglobin <13.5 g/dL for men and <12.0 g/dL for women.
* Postmenopausal
* Smoking
* Use of chronic Medications (aspirin, statins, anti-inflammatory drugs)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2012-11; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Change in Brachial artery diameter in response to hyperemia. | Baseline and 15 min after hyperemia
  Endothelial function test - Arterial endothelial function will be assessed non-invasively by ultrasound examination of the arterial endothelium dependent vasodilation response to reactive hyperemia. The right brachial artery, proximal to the antecubital fossa, will be imaged longitudinally using a linear-array transducer. Flow-mediated endothelium-dependent vasodilation will be assessed by measuring the brachial artery diameter at baseline and during reactive hyperemia. Reactive hyperemia will be induced by deflating a cuff previously inflated to 200 mmHg for 5 minutes in the forearm. Variables will be measured for three consecutive cardiac cycles and the average will be taken.

CONTACTS AND LOCATIONS:
Overall Officials: Virend K Somers, MD PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States